CLINICAL TRIAL: NCT06063603
Title: Pilot Test of a Pain Management Intervention Preparatory to a Future Pragmatic Trial (ASCENT)
Brief Title: Evaluation of a Pain Management Intervention Preparatory to a Future Pragmatic Trial, ASCENT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ASCENT_Pilot; NCI-2023-05223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ASCENT (Other: Mayo Clinic in Rochester); 23-004139 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-09-13; First posted 2023-10-02 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Leukemia; Hematopoietic and Lymphoid System Neoplasm; Lymphoma; Malignant Solid Neoplasm; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Acupuncture Therapy; Cognitive Behavioral Therapy; Early Intervention, Educational; Educational Status; Methods; Exercise; Exercise Therapy; Interviews as Topic; Massage; Mindfulness; Mindfulness-Based Stress Reduction; Analgesia; Pain Management; Palliative Care; Patient Comfort; Patient Navigation; Referral and Consultation; Spiritual Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Pain management) (Experimental): See detailed description.
  Interventions: Procedure: Acupuncture Therapy; Behavioral: Cancer Pain Management; Behavioral: Cognitive Behavior Therapy; Other: Educational Intervention; Other: Exercise; Other: Interview; Procedure: Massage Therapy; Behavioral: Mindfulness Relaxation; Procedure: Pain Therapy; Other: Palliative Therapy; Behavioral: Patient Navigation; Other: Referral; Procedure: Spiritual Therapy; Procedure: Spiritual Care Referral; Other: Survey Administration
- Group II (Interview) (Active Comparator): ASCENT study interventionists complete an interview on study.
  Interventions: Other: Interview
- Group III (Focus group) (Active Comparator): Medical oncology providers participate in a focus group on study.
  Interventions: Procedure: Discussion

INTERVENTIONS:
Procedure: Acupuncture Therapy — Undergo acupuncture therapy
  Other Names: Acupuncture
  Arms: Group I (Pain management)
Behavioral: Cancer Pain Management — Receive pain clinic referral
  Other Names: management of cancer pain
  Arms: Group I (Pain management)
Behavioral: Cognitive Behavior Therapy — Undergo CBT
  Other Names: CBT; cognitive therapy; CT
  Arms: Group I (Pain management)
Procedure: Discussion — Participate in focus group
  Other Names: Discuss
  Arms: Group III (Focus group)
Other: Educational Intervention — Receive self-guided pain management education materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (Pain management)
Other: Exercise — Participate in exercise
  Other Names: Exercise Type
  Arms: Group I (Pain management)
Other: Interview — Complete interview
  Arms: Group I (Pain management); Group II (Interview)
Procedure: Massage Therapy — Receive massage
  Other Names: Massage
  Arms: Group I (Pain management)
Behavioral: Mindfulness Relaxation — Practice mindfulness
  Other Names: MBSR; Mindful Meditation; Mindfulness Meditation; Mindfulness-Based Stress Reduction
  Arms: Group I (Pain management)
Procedure: Pain Therapy — Receive pain treatment/medicine
  Other Names: Analgesia; Pain Control; Pain Management; Pain, Pain Management
  Arms: Group I (Pain management)
Other: Palliative Therapy — Receive palliative care referral
  Other Names: Comfort Care; PA-Palliative Therapy; palliation; Palliative; Palliative Care; Palliative Treatment; Symptom Management; Symptoms Management
  Arms: Group I (Pain management)
Behavioral: Patient Navigation — Undergo visits with PCM and CHW for pain management
  Other Names: Patient Navigator Program
  Arms: Group I (Pain management)
Other: Referral — Receive pain management referrals
  Other Names: Referred
  Arms: Group I (Pain management)
Procedure: Spiritual Therapy — Receive spiritual support
  Arms: Group I (Pain management)
Procedure: Spiritual Care Referral — Receive spiritual care referral
  Arms: Group I (Pain management)
Other: Survey Administration — Ancillary studies
  Arms: Group I (Pain management)

SUMMARY:
This clinical trial tests how well a pain management intervention preparatory to a future pragmatic trial works in rural dwelling and Hispanic cancer survivors. Cancer pain is a key case study in health disparities in the United States. Cancer pain is prevalent, under treated, and remains a major cause of suffering, impairment, and disability for millions of Americans. Individual pain interventions and care models show promise for cancer pain in controlled settings. Hispanic and rural-dwelling cancer survivors stand to benefit the most from electronic health record innovations, as each of these health disparities populations experience profound disparities in pain outcomes, including marked under- and over-prescribing of opioids. Additionally, Hispanics not only comprise a steadily growing proportion of cancer survivors, but are also increasingly immigrating to rural communities, potentially placing them at "double risk" for poor outcomes. This trial will allow for the refinement of pain management intervention components that could help the management of cancer-related pain in rural dwelling and Hispanic cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To refine and pilot test components of a validated collaborative care model-based intervention aimed at improving pain control among rural dwelling and Hispanic cancer survivors.

GROUP I: Participants meet with pain care manager (PCM) and community health worker (CHW) via telephone or video visit to discuss the cancer-related pain. Participants receive self-guided pain management education materials and receive an action plan with suggestions or referrals to participate in tier 1 interventions that include exercise, cognitive behavioral therapy, medication and/or tier 2 interventions that include integrative medicine (massage, acupuncture and mindfulness relaxation), spiritual support, pain clinic referral and palliative and spiritual care referrals during the intake visit. Participants undergo a planning visit 2 weeks later to give an update on their pain and may receive additional resources from the PCM and/or CHW. Participants then undergo a final visit 4 weeks later with the PCM and/or CHW and receive final recommendations and referrals. Participants may receive a follow up call between intake and visit 2 and/or between visit 2 and the final visit from the CHW or PCM to assess pain levels on study.

GROUP II: ASCENT study interventionists complete an interview on study.

GROUP III: Medical oncology providers participate in a focus group on study.

ELIGIBILITY:
Inclusion Criteria:

* A qualifying liquid or solid cancer diagnosis with visits at a participating Mayo site
* Age 18+
* Numerical rating scale (NRS) pain score of a 5+ out of 10
* Pain that developed (onset) or significantly worsened since cancer diagnosis
* Malignant hematology including:

  * Lymphoma
  * Myeloma
  * Chronic leukemias

Exclusion Criteria:

* Patient Health Questionnaire (PHQ) 8 score of 10 or more
* Life expectancy less than 12 months
* Hospice enrollment
* Admitted to hospital from long term care/skilled nursing facilities (SNF)
* Acute leukemias
* Primary brain tumors
* Confinement to a bed or a chair more than a third of waking hours because of health complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L. Cheville, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only Group 1 were actual participants who were enrolled in the study and received the intervention. Data was only collected for Group 1, so this is the only data reported.
  Group 2 consisted of interventionalists (provided the intervention to Group 1 participants). Group 3 were Medical Oncology providers. Neither Group 2 nor 3 received any intervention or were enrolled in the study. Groups 2 and 3 participated only in study development.
Groups:
- Group I (Pain Management): See detailed description.
  Acupuncture Therapy: Undergo acupuncture therapy
  Cancer Pain Management: Receive pain clinic referral
  Cognitive Behavior Therapy(CBT): Undergo CBT
  Educational Intervention: Receive self-guided pain management education materials
  Exercise: Participate in exercise
  Interview: Complete interview
  Massage Therapy: Receive massage
  Mindfulness Relaxation: Practice mindfulness
  Pain Therapy: Receive pain treatment/medicine
  Palliative Therapy: Receive palliative care referral
  Patient Navigation: Undergo visits with pain care manager (PCM) and community health worker (CHW) for pain management
  Referral: Receive pain management referrals
  Spiritual Therapy: Receive spiritual support
  Spiritual Care Referral: Receive spiritual care referral
  Survey Administration: Ancillary studies
- Group 2 (Intervention Providers): Study interventionalists complete an interview on study.
- Group 3 (Medical Oncology Providers): Medical oncology providers participate in a focus group on study.
Period: Overall Study
Arm/Group | Group I (Pain Management) | Group 2 (Intervention Providers) | Group 3 (Medical Oncology Providers)
Started | 51 | 5 | 3
Completed Intake Visit | 44 | 0 | 0
Completed Planning Visit | 43 | 0 | 0
Completed Final Visit | 41 | 0 | 0
Completed Survey | 35 | 0 | 0
Participated in Focus Group | 0 | 0 | 3
Participated in Interventionalist's Interview | 0 | 5 | 0
Completed | 35 | 5 | 3
Not Completed | 16 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Groups II and III were not enrolled to the study. They participated in development and evaluation of this pilot as providers. These groups did not receive the study intervention, and no demographic or outcome data was collected from these groups. Only data from Group 1 is reported.
Arm/Group | Group I (Pain Management)
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.03922 (12.69167)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 51
Rural-Urban Commuting Area (RUCA) category [Count of Participants; unit: Participants]
  Urban (RUCA 1-3) | 18
  Large rural (RUCA 4-6) | 1
  Small rural (RUCA 7-9) | 3
  Rural (RUCA 10) | 29
Cancer type [Count of Participants; unit: Participants]
  Breast | 13
  Endocrine | 2
  GI | 7
  GYN | 1
  Genitourinary | 4
  Head and neck | 2
  Heme | 9
  Lung | 5
  Melanoma | 2
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention
Description: Assessed by proportion of participants who received key intervention components.
Time Frame: Up to 60 days
Population: Participants who completed all three visits were sent a survey about their experience with the ASCENT pilot--of the 41 who completed all 3 visits, 35 completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pain Management)
Number analyzed (Participants) | 51
Participants
  Completed intake visit, planning visit, and final visit | 41
  Utilized materials sent to the portal: number analyzed (Participants) | 35
  Utilized materials sent to the portal | 17
  Utilized mailed materials that discussed pain management techniques: number analyzed (Participants) | 35
  Utilized mailed materials that discussed pain management techniques | 11
  Utilized ASCENT website: number analyzed (Participants) | 35
  Utilized ASCENT website | 5
  Utilized follow-up phone calls with a member of the ASCENT team: number analyzed (Participants) | 35
  Utilized follow-up phone calls with a member of the ASCENT team | 27
  Utilized the Action Plan: number analyzed (Participants) | 35
  Utilized the Action Plan | 16

2. Primary Outcome: Acceptability of Intervention - Interaction
Description: As assessed by frequency of participant interaction with care team.
Time Frame: Up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pain Management)
Number analyzed (Participants) | 35
Participants
  Never | 0
  Once | 1
  Every other week | 18
  Weekly | 16
  Multiple times a week | 0

3. Primary Outcome: Acceptability of Intervention - Satisfaction
Description: As assessed by participant satisfaction with care team interactions
Time Frame: Up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pain Management)
Number analyzed (Participants) | 35
Participants
  Not satisfied with frequency of communication with a member of the ASCENT care team | 0
  Satisfied with frequency of communication with a member of the ASCENT care team | 35

4. Primary Outcome: Utility of Intervention - Helpfulness
Description: Assessed by study-specific questionnaire. Questions were answered on an Adjectival Ordinal 5-point scale where 1 = not at all and 5 = extremely helpful.
Time Frame: Up to 60 days
Population: Participants were asked about the helpfulness of specific components of the ASCENT intervention if and only if they utilized that component.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pain Management)
Number analyzed (Participants) | 35
Participants
  Helpfulness of working with the ASCENT care team: Not at all helpful | 2
  Helpfulness of working with the ASCENT care team: Somewhat helpful | 7
  Helpfulness of working with the ASCENT care team: Helpful | 6
  Helpfulness of working with the ASCENT care team: Very helpful | 9
  Helpfulness of working with the ASCENT care team: Extremely helpful | 11
  Helpfulness of the materials sent to the patient portal: number analyzed (Participants) | 17
  Helpfulness of the materials sent to the patient portal: Not at all helpful | 0
  Helpfulness of the materials sent to the patient portal: Somewhat helpful | 1
  Helpfulness of the materials sent to the patient portal: Helpful | 4
  Helpfulness of the materials sent to the patient portal: Very helpful | 8
  Helpfulness of the materials sent to the patient portal: Extremely helpful | 4
  Helpfulness of the mailed materials that discussed different pain management techniques: number analyzed (Participants) | 11
  Helpfulness of the mailed materials that discussed different pain management techniques: Not at all helpful | 0
  Helpfulness of the mailed materials that discussed different pain management techniques: Somewhat helpful | 1
  Helpfulness of the mailed materials that discussed different pain management techniques: Helpful | 4
  Helpfulness of the mailed materials that discussed different pain management techniques: Very helpful | 5
  Helpfulness of the mailed materials that discussed different pain management techniques: Extremely helpful | 1
  Helpfulness of the ASCENT website: number analyzed (Participants) | 5
  Helpfulness of the ASCENT website: Not at all helpful | 0
  Helpfulness of the ASCENT website: Somewhat helpful | 0
  Helpfulness of the ASCENT website: Helpful | 2
  Helpfulness of the ASCENT website: Very helpful | 0
  Helpfulness of the ASCENT website: Extremely helpful | 3
  Helpfulness of the follow-up phone calls with a member of the ASCENT team: number analyzed (Participants) | 27
  Helpfulness of the follow-up phone calls with a member of the ASCENT team: Not at all helpful | 0
  Helpfulness of the follow-up phone calls with a member of the ASCENT team: Somewhat helpful | 4
  Helpfulness of the follow-up phone calls with a member of the ASCENT team: Helpful | 3
  Helpfulness of the follow-up phone calls with a member of the ASCENT team: Very helpful | 11
  Helpfulness of the follow-up phone calls with a member of the ASCENT team: Extremely helpful | 9
  Helpfulness of the Action Plan: number analyzed (Participants) | 16
  Helpfulness of the Action Plan: Not at all helpful | 0
  Helpfulness of the Action Plan: Somewhat helpful | 1
  Helpfulness of the Action Plan: Helpful | 3
  Helpfulness of the Action Plan: Very helpful | 4
  Helpfulness of the Action Plan: Extremely helpful | 8

5. Primary Outcome: Utility of Intervention - Confidence
Description: Assessed by study-specific questionnaire. Questions were answered on an Adjectival Ordinal 5-point scale where 1 = not at all confident and 5 = extremely confident.
Time Frame: Up to 60 days
Population: Five patients did not set goals and thus the question about setting goals with the care team was not applicable.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pain Management)
Number analyzed (Participants) | 35
Participants
  Confidence in achieving goal(s) set with the ASCENT care team as part of the action plan: Not at all confident | 2
  Confidence in achieving goal(s) set with the ASCENT care team as part of the action plan: Somewhat confident | 3
  Confidence in achieving goal(s) set with the ASCENT care team as part of the action plan: Confident | 6
  Confidence in achieving goal(s) set with the ASCENT care team as part of the action plan: Very confident | 10
  Confidence in achieving goal(s) set with the ASCENT care team as part of the action plan: Extremely confident | 9
  Confidence in achieving goal(s) set with the ASCENT care team as part of the action plan: N/A | 5
  Confidence in ability to find resources to help with pain: Not at all confident | 6
  Confidence in ability to find resources to help with pain: Somewhat confident | 7
  Confidence in ability to find resources to help with pain: Confident | 6
  Confidence in ability to find resources to help with pain: Very confident | 13
  Confidence in ability to find resources to help with pain: Extremely confident | 3
  Confidence in ability to find resources to help with pain: N/A | 0
  Confidence in managing pain better in the future: Not at all confident | 5
  Confidence in managing pain better in the future: Somewhat confident | 9
  Confidence in managing pain better in the future: Confident | 5
  Confidence in managing pain better in the future: Very confident | 13
  Confidence in managing pain better in the future: Extremely confident | 3
  Confidence in managing pain better in the future: N/A | 0

6. Primary Outcome: Utility of Intervention - Ease
Description: Assessed by study-specific questionnaire. Questions were answered on an Adjectival Ordinal 5-point scale where 1 = very difficult and 5 = extremely easy.
Time Frame: Up to 60 days
Population: Participants were asked about the ease of use of specific components of the ASCENT intervention if and only if they utilized these components. Five participants did not utilize these components.
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Pain Management)
Number analyzed (Participants) | 35
Participants
  Ease of understanding materials sent to the patient portal: number analyzed (Participants) | 17
  Ease of understanding materials sent to the patient portal: Very difficult | 0
  Ease of understanding materials sent to the patient portal: Somewhat difficult | 0
  Ease of understanding materials sent to the patient portal: Neither easy nor difficult | 0
  Ease of understanding materials sent to the patient portal: Somewhat easy | 2
  Ease of understanding materials sent to the patient portal: Very easy | 15
  Ease of understanding mailed materials that discussed pain management techniques: number analyzed (Participants) | 11
  Ease of understanding mailed materials that discussed pain management techniques: Very difficult | 0
  Ease of understanding mailed materials that discussed pain management techniques: Somewhat difficult | 0
  Ease of understanding mailed materials that discussed pain management techniques: Neither easy nor difficult | 1
  Ease of understanding mailed materials that discussed pain management techniques: Somewhat easy | 2
  Ease of understanding mailed materials that discussed pain management techniques: Very easy | 8
  Ease of understanding the ASCENT website: number analyzed (Participants) | 5
  Ease of understanding the ASCENT website: Very difficult | 0
  Ease of understanding the ASCENT website: Somewhat difficult | 0
  Ease of understanding the ASCENT website: Neither easy nor difficult | 0
  Ease of understanding the ASCENT website: Somewhat easy | 2
  Ease of understanding the ASCENT website: Very easy | 3
  Ease of understanding follow-up phone calls with a member of the ASCENT team: number analyzed (Participants) | 27
  Ease of understanding follow-up phone calls with a member of the ASCENT team: Very difficult | 0
  Ease of understanding follow-up phone calls with a member of the ASCENT team: Somewhat difficult | 0
  Ease of understanding follow-up phone calls with a member of the ASCENT team: Neither easy nor difficult | 2
  Ease of understanding follow-up phone calls with a member of the ASCENT team: Somewhat easy | 1
  Ease of understanding follow-up phone calls with a member of the ASCENT team: Very easy | 24
  Ease of understanding the Action Plan: number analyzed (Participants) | 16
  Ease of understanding the Action Plan: Very difficult | 0
  Ease of understanding the Action Plan: Somewhat difficult | 0
  Ease of understanding the Action Plan: Neither easy nor difficult | 1
  Ease of understanding the Action Plan: Somewhat easy | 0
  Ease of understanding the Action Plan: Very easy | 15

ADVERSE EVENTS:
Time Frame: Up to 60 days
Description: Groups II and III did not participate in the intervention and were not enrolled to the study. Adverse events were not collected from the provider and interventionalist participants in Group II or III.
Groups:
- Group II (Intervention Providers): Group II participants were not enrolled to the study and participated only in study development.
- Group III (Medical Oncology Providers): Group III participants were not enrolled to the study and participated only in study development.
Arm/Group | Group I (Pain Management) | Group II (Intervention Providers) | Group III (Medical Oncology Providers)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/51 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT06063603/Prot_SAP_000.pdf